CLINICAL TRIAL: NCT03330730
Title: A Randomized, Controlled, Multicenter, Prospective, Open Study Evaluating the Efficiency of the IsereADOM Home-care Service Package in the Prevention of Unplanned Hospitalizations of Patients With Cancer
Brief Title: Evaluation of the Efficiency of the IsereADOM Home-care Service Package in the Prevention of Unplanned Hospitalizations of Patients With Cancer
Acronym: IsereADOM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Leon Berard (Other)
Collaborators: Conseil general de l'Isere (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: IsereADOM
Record Dates: First submitted 2017-10-25; First posted 2017-11-06 (Actual); Last update posted 2019-12-13 (Actual); Status verified 2019-12

CONDITIONS: Neoplasms
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental (Experimental): Patients with oncological follow up and home-care service package IsereADOM:
  Objects connected to patients' home (thermometer, weight scale, tensiometer +/- oximeter, glucose meter or pedometer) with graduated protocol for medical platform support.
  Digital linkbook (different from the medical file) accessible to the patient and the standard care actors.
  Referent sentinel: a field actor to coordinate the care. Preferred contact of the patient outside the center Motivational coaching: 1 to 2 axes to be defined by the investigator among the following axes (physical activity, nutrition and hydration, drug compliance, medical follow-up, chronic and moral pain, acceptance of the disease and treatments).
  Interventions: Other: IsereADOM service package
- Control (No Intervention): Patients with oncological follow up only

INTERVENTIONS:
Other: IsereADOM service package — Objects connected to patients' homes (thermometer, weight scale, tensiometer +/- oximeter, glucose meter or pedometer), Digital liaison booklet, Sentinel referent, Motivational coaching
  Arms: Experimental

SUMMARY:
The main objective of the project is to compare the effectiveness and efficiency of innovative care through the IsereADOM home-care service package versus standard care in the prevention of unplanned hospitalizations in patients with cancer treatment. In accordance with the recommendations of the French High Authority of Health (HAS), a cost-utility analysis (ACU) will be implemented

DETAILED DESCRIPTION:
Specific management of cancer patients involves carrying out often heavy treatments (surgery, chemotherapy, radiotherapy, interventional radiology, etc.) during which close coaching is necessary. In spite of this adapted follow-up, the natural evolution of the disease and the management of treatment tolerance make these patients a frail population, sometimes isolated, for which admission to emergency services and admission to full hospitalization can be required.

This trial will use a service package at home named IsereADOM, currently in the development phase in the management of 4 types of populations:

* Retired persons with no proven loss of autonomy;
* Users with loss of autonomy at risk of falling;
* Cardiac insufficiency;
* Patients with cancer.

This service package is based on the identification of a person of proximity, called "sentinel referent". This person, in charge of monitoring the patient at his / her home, has access to various connected tools installed at the patient's home (scales, tensiometer ...) as well as computer solutions enabling the sharing of information with the different actors in the management of the patient.

In addition, the patient benefits from motivational coaching based on investigator's recommendation and telephone and internet information platforms.

ELIGIBILITY:
Inclusion Criteria:

* age > or = 18 years old at the time of signature of informed consent form
* patient with solid or hematologic tumor under treatment for cancer at the time of inclusion
* Patient managed in a medical emergency context in the 2 weeks prior to inclusion
* Patient living in Isère department (area of coverage of experiment)
* ECOG Performance index < or = 3
* patient with a life expectancy of 6 months or more
* patient with social security system
* patient able to read, write and understand French
* patient with signed informed consent

Exclusion Criteria:

* Patient included in clinical trial evaluating early stage therapeutic innovation with pharmacokinetic sampling
* Patients with follow-up in Hospitalization at Home at the end of the hospitalization for inclusion
* Patient without help "referent" in the entourage (spouse, family, friend ...)
* Patient residing in Elderly Accommodation (EHPAD) or in any other institution for dependent persons
* Patient who is homeless or living in a home that does not allow the installation of the necessary equipment
* Patient with severe cognitive impairment, defined by score at Mini Mental State Examination (MMSE)< 23/30
* Patient unable to comply (or unwilling to comply) with follow-up of the study for the duration of participation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2018-01-11 (Actual); Primary Completion 2019-06-17 (Actual); Study Completion 2019-06-17 (Actual)

PRIMARY OUTCOMES:
Comparison of the effectiveness and efficiency of innovative care with the IsereADOM home-care service package versus standard support | 6 months
  Comparison of the mean number of unplanned hospitalizations observed within 6 months of randomization.
Incremental Cost-Utility Ratio comparison | 6 months
  Evaluation of the costs of the home-care service package; Assessment of health care consumption from a community perspective; Calculation of the years of life gained in good health (QALY)

SECONDARY OUTCOMES:
Budget impact analysis | 6 months
  Calculation of incremental costs and saved costs with the experimental strategy
Patient's condition evaluation | 6 months
  Evaluation in both arms of loss of autonomy with questionnaires "Activities of Daily Living"
Patient's condition evaluation | 6 months
  Evaluation in both arms of loss of autonomy with questionnaires "Instrumental Activities of Daily Living"
Patient's condition evaluation | 6 months
  Evaluation in both arms of anxiety with questionnaire "Hospital Anxiety and Depression scale"
Patient's condition evaluation | 6 months
  Evaluation in both arms of depression with questionnaire "Hospital Anxiety and Depression scale"
Patient's condition evaluation | 6 months
  Evaluation in both arms of nutritional status by measuring albumin rate
Patient's condition evaluation | 6 months
  Evaluation in both arms of nutritional status by measuring prealbumin rate
Patient's condition evaluation | 6 months
  Evaluation in both arms of nutritional status by measuring weight
Patient's condition evaluation | 6 months
  Evaluation in both arms of the quality of life with questionnaire "EuroQoL 5 Dimensions 5 Levels"
Patient's condition evaluation | 6 months
  Description in both arms of home care with questionnaire "RUD" for the natural caregivers
Patient's condition evaluation | 6 months
  Evaluation in both arms of consumption of unprogrammed care with patient's booklet
Patient's condition evaluation | 6 months
  Evaluation in both arms of overall survival
Patient's condition evaluation | 6 months
  Characterizing unjustified hospitalizations, to determine predictive factors for the efficiency of experimental management, progression-Free Survival
Evaluation of IsereADOM home-care service package impact | 6 months
  Evaluation of the duration of setting up the experimental procedure by measuring the delay between the randomisation and the complete installation of the home-care service package at the patient's home
Evaluation of IsereADOM home-care service package impact | 6 months
  Evaluation of the proportion of sentinel nurses asked to participate in the study
Evaluation of IsereADOM home-care service package impact | 6 months
  Evaluation of the number of calls and the number of connections to the telephone and Internet platforms
Evaluation of IsereADOM home-care service package impact | 6 months
  Evaluation of the number of refusal to participate.
Evaluation of IsereADOM home-care service package impact | 6 months
  Evaluation of the causes of refusal to participate.
Analysis of the geographical factors predicting the effectiveness of the package | 6 months

CONTACTS AND LOCATIONS:
Locations (3):
- France (3):
  - Centre Léon Bérard, Lyon, Auvergne-Rhône-Alpes
  - CHU Grenoble Alpes, Grenoble
  - Institut Daniel Hollard, Grenoble